CLINICAL TRIAL: NCT04528771
Title: Proof of Concept Safety Trial for S-Nitrosylation Therapy to Improve Oxygenation Status in Severe Covid-19 Patients Receiving Supplemental Oxygen Support
Brief Title: S-Nitrosylation Therapy of COVID-19
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study delays
Sponsor: James Reynolds (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor-Investigator, James Reynolds, Principal Investigator, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY20210599
Record Dates: First submitted 2020-08-25; First posted 2020-08-27 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV2 Infection; Covid19
Keywords: respiratory distress; respiratory failure
MeSH Terms: conditions — COVID-19; Dyspnea; Respiratory Insufficiency | interventions — Nitrogen

STUDY DESIGN:
Intervention Model Description: Single-site, double-blinded, randomized, placebo controlled trial with a superiority design. The study will randomize 24 patients 1:1 (12 treatment vs 12 control) to either S-nitrosylation therapy or placebo arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational product will be prepared and dispensed by designated unblinded site personnel at the pharmacy; the investigational product label will indicate the study number but will not indicate the treatment assignment. Any site personnel involved in the administration and assessment of the investigational product will be blinded to subject treatment assignments throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SNO (Experimental): 12 patients in the S-nitrosylation arm will receive SNO (six-hour treatment with a sequential increasing dose regimen of 20 ppm x 2 hr, 40 ppm x 2 hr, 80 ppm x 2 hr).
  Interventions: Drug: SNO
- Placebo (Placebo Comparator): 12 patients in the placebo arm will receive nitrogen gas (six-hour treatment).
  Interventions: Drug: Nitrogen gas

INTERVENTIONS:
Drug: SNO — Six-hour SNO treatment by inhalation at a sequential increasing dose regimen of 20 ppm x 2 hr, 40 ppm x 2 hr, 80 ppm x 2 hr. Patient care and follow-up during and after ENO administration will follow the critical care clinical SOPs developed by our institution (attached in Additional Information), which are consistent with the guidelines set out by the World Health Organization.
  Arms: SNO
Drug: Nitrogen gas — Six-hour nitrogen gas treatment by inhalation.Patient care and follow-up during and after ENO administration will follow the critical care clinical SOPs developed by our institution (attached in Additional Information), which are consistent with the guidelines set out by the World Health Organization.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to provide expanded access of S-nitrosylation therapy for the treatment of severe acute respiratory syndrome coronavirus (SARS-CoV2) infection.

DETAILED DESCRIPTION:
Randomized controlled trial for safety of a 6-hour escalating dose of S-nitrosylation therapy or placebo to ventilated patients. This will be a single-site study conducted within the UH-CMC medical ICU designated COVID-19 quarantine areas.

ELIGIBILITY:
Inclusion Criteria (Severe COVID-19 Status)

* Hospitalized with confirmed SARS-CoV-2 infection by polymerase chain reaction (PCR) or other validated tests as they become available within 30 days of enrollment.
* In mild respiratory distress, defined as a P/F ratio of between 200 and 325 mm Hg.
* Spontaneously breathing subjects receiving > 4 liters/min of oxygen.
* Patients enrolled and able to start ENO treatment after oxygen stabilization.
* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent, or enrolled under International Conference on Harmonization (ICH) E6(R2) 4.8.15 emergency use provisions as deemed necessary by the investigator (participants ≥ 18 years of age).
* 18-89 years of age

Exclusion Criteria

* COVID-19 patients with mild to no respiratory distress, defined as P/F ratio > 325 mm Hg.
* COVID-19 patients receiving supplemental oxygen equivalent to an FiO2 of > 0.90 (reduction of FiO2 at this level or higher when ENO is blended into gas source cannot be avoided).
* COVID-19 patients receiving supplemental oxygen with active ventilatory support, CPAP, etc.
* Physician of record opposed to enrolling the patient due to perceived safety concerns; or any condition that does not allow the protocol to be followed safely.
* Subjects with past medical history of lung malignancy or pneumonectomy or lung transplant
* Subjects who have a history of malignancy or other irreversible disease/conditions with a 6-month mortality > 50%
* Subjects that have experienced cardiac arrest with CPR for longer than 30 minutes
* Patients on extracorporeal membrane oxygenation (ECMO) + patients intubated on ventilator
* Patient groups at an increased risk to form methemoglobin. (e.g. congenital variants of Met-Hb)
* Patients with anemia, defined as a hemoglobin of < 9 g/dL
* Individuals who are pregnant or breastfeeding
* Individuals with an acute disorder or history of chronic diseases of the heart, lungs, kidney, liver, or any other medical condition that in the opinion of the screening physician makes them unsuitable for study.
* Individuals taking nitrates.
* Individuals receiving PDE-5 inhibitors, any drugs that are nitric oxide donors (e.g. prilocaine, sodium nitroprusside and nitroglycerine), drugs known to increase methemoglobin (e.g. lidocaine, prilocaine, benzocaine, or dapsone), drugs that interfere with nitrite metabolism (e.g. allopurinol) and drugs that may potentiate hypotension (e.g. antihypertensives, diuretics, meperidine).
* Individuals with an inherited or acquired blood coagulation disorder, congenital methemoglobinemia, or a familial hemoglobinopathy that impacts oxygen delivery (e.g. sickle cell).
* Individuals who might have difficulty with the placement of a face mask (e.g. claustrophobia, uncontrolled asthma, severe allergies, sensitive skin) and/or the inhalation of a product for approximately 6 hours.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | 30 days
  Adverse events related to SNO therapy.
Frequency of Intubation | 30 days
  Number of intubations required.
Progression to use of ECMO | 30 days
  Use of ECMO required.

SECONDARY OUTCOMES:
Time to Clinical Status Improvement | 30 days
  Number of days required to see a greater than or equal to 2 point improvement on the WHO 9-point clinical status assessment ordinal scale.
  Clinical status will be assessed using the WHO 9-point ordinal scale as follows:
  0. Uninfected - no clinical or virological evidence of infection
  1. Ambulatory - no limitation of activities
  2. Ambulatory - Limitation of activities
  3. Hospitalized, mild disease - no oxygen therapy
  4. Hospitalized, mild disease - oxygen by mask or nasal prongs
  5. Hospitalized, severe disease - non-invasive ventilation or high-flow oxygen
  6. Hospitalized, severe disease - intubation and mechanical ventilation
  7. Hospitalized, severe disease - ventilation + additional organ support (pressors, RRT, ECMO)
  8. Dead
Clinical Status | 30 days
  Proportion of patients in each stage at maximum severity on the 9-point clinical status assessment ordinal scale.
  Clinical status will be assessed using the WHO 9-point ordinal scale as follows:
  0. Uninfected - no clinical or virological evidence of infection
  1. Ambulatory - no limitation of activities
  2. Ambulatory - Limitation of activities
  3. Hospitalized, mild disease - no oxygen therapy
  4. Hospitalized, mild disease - oxygen by mask or nasal prongs
  5. Hospitalized, severe disease - non-invasive ventilation or high-flow oxygen
  6. Hospitalized, severe disease - intubation and mechanical ventilation
  7. Hospitalized, severe disease - ventilation + additional organ support (pressors, RRT, ECMO)
  8. Dead
Respiratory Clinical Status | 30 days
  Respiratory clinical status assessed by a 7-point respiratory status ordinal scale that captures oxygen requirement, ventilator support or death.
  7-Point Respiratory Severity Scale Range: 1-7 Higher values = worse
  1. Not receiving oxygen supplementation; AND room air oxygen saturation ≥ 95%
  2. Supplemental oxygen ≤ 2 liters/min; OR room air oxygen saturation ≤ 94%
  3. Supplemental nasal oxygen >2 and <= 5 liters/min
  4. Supplemental nasal oxygen >5 liters/min
  5. HFNC or NIV with FiO2 > 50%
  6. Intubation or ECMO
  7. Death
Duration of Hospitalization | 30 days
  Duration of total hospitalization days as measured by total hospitalization, ventilator and ICU days
All-Cause Mortality | 30, 60 days
  All-cause mortality
Time to Discontinuation of Oxygen Therapy | 30 days
  Number of days required to discontinue oxygen supportive therapy
Discontinuation of Oxygen Therapy | 30 days
  Proportion of patients alive and with discontinued oxygen supportive therapy at day 30

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schilz, DO, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States